CLINICAL TRIAL: NCT06037161
Title: Comparison of Surgical Techniques to Treat Isolated Gingival Recession in Mandibular Incisors: A Randomized Clinical Trial
Brief Title: Comparison of Two Methods of Covering a Single Lower Front Tooth With Receded Gums
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Case Western Reserve University (Other)
Responsible Party: Principal Investigator, Gian Schincaglia, Professor, Chair and Graduate Program Director, Case Western Reserve University
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY20220902
Record Dates: First submitted 2023-08-30; First posted 2023-09-14 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Recession, Gingival
Keywords: Connective tissue graft(s); cosmetic periodontal plastic surgery; gingival recession; mucogingival surgery; treatment planning
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GPST + CTG (Experimental): Gingival Pedicle Split Thickness + Connective Tissue Graft procedure
  Interventions: Procedure: Mandibular Incisor root coverage procedure
- CAF + CTG (Active Comparator): Coronally Advanced Flap + Connective Tissue Graft procedure
  Interventions: Procedure: Mandibular Incisor root coverage procedure

INTERVENTIONS:
Procedure: Mandibular Incisor root coverage procedure — Mucogingival procedure to cover mandibular incisor tooth with receded gums

SUMMARY:
The primary objective of this randomized clinical trial is to compare the mean root coverage achieved with Coronally Advanced Flap (CAF) + Connective Tissue Graft (CTG) (control) to Gingival Pedicle Split Thickness flap (GPST) + CTG (test) for the treatment of isolated gingival recession defects in mandibular incisors. The secondary objectives are to compare the percentage of complete root coverage and keratinized tissue gain between the two techniques.

DETAILED DESCRIPTION:
1. Research Scope: This study focuses on treatment of isolated gingival recession in mandibular incisors. Coronally advanced flap (CAF) with connective tissue graft (CTG) is the most predictable surgical technique for recession coverage (Chambrone and Tatakis 2015). However the early data indicate that CAF+CTG provides low predictability of root coverage of recessions in mandibular incisors (Zucchelli et al. 2014). We recently described a surgical technique called gingival pedicle split-thickness tunnel (GPST)+CTG. This technique entails a modified flap design to maximize recession coverage in mandibular incisors (Agusto et al 2019). The preliminary data using GPST+CTG shows complete root coverage in 98% of the treated sites (Schincaglia et al.2022). This study will compare CAF+CTG versus GPST+CTG for the management of isolated gingival recession in mandibular incisors. Clinical measurements will be performed at baseline and 6-months after the surgery to study the difference in results achieved by these two surgical techniques.
2. Objectives: The primary objective of this randomized clinical trial is to compare the mean root coverage achieved with CAF+CTG (control) to GPST+CTG (test) for the treatment of isolated gingival recession defects in mandibular incisors. The secondary objectives are to compare the percentage of complete root coverage and keratinized tissue gain between the two techniques.
3. Hypothesis: It is predicted that the GPST+CTG technique will be superior to CAF+CTG in terms of mean root coverage, complete root coverage and keratinized tissue gain at 6-months post-surgery.
4. Justification for the proposal: Although subepithelial connective tissue graft is considered the gold standard approach for the management of gingival recessions (Chambrone and Tatakis 2015; Greenwell et al. 2005), data indicates lower efficacy of CAF+CTG in the treatment of isolated gingival recession in mandibular incisors. Anatomical challenges in this area such as muscular tension, high labial frenum insertion, limited tissue thickness and vestibular depth seem to reduce the predictability of the procedure (Zucchelli et al. 2014). The use of a modified flap design (GPST) in combination with CTG was introduced by our group to treat isolated advanced gingival recession in mandibular incisors. This technique seems to provide a higher success rate for root coverage in this specific clinical condition. A predictable technique for the treatment of isolated recession defects in mandibular incisors is needed since gingival recessions on mandibular incisors represent 42% of the total prevalence of recessions in the general population (Mythri et al. 2015). In addition, a technique that provides high predictability for root coverage will eliminate or minimize the need for revision surgical procedures. A revision surgery is performed when the first surgical procedure did not achieve the desired clinical results. Eliminating the need of a revision procedure will save time for the clinician and will eliminate pain and discomfort of an additional surgical procedure to the patient.

This study will be conducted as a single-blinded, randomized controlled clinical trial in accordance with the CONSORT guidelines (Moher et al., 2012). Upon approval of the partial HIPAA waiver, pre-screening will take place through a phone questionnaire for subjects recruited through flyers and social media to assess for preliminary eligibility. The study will include the following phases: 1. Screening and recruiting 2. Initial therapy, baseline clinical measurements 3. Surgical therapy 4. Post-operative follow-up at 2-, 6-weeks 5. Clinical measurements at 6-months after surgery. Screening and recruiting: Upon consenting, screening will include gathering patient's personal information, medical history through questionnaires and clinical examination to confirm eligibility. Medical consultation with the patient's physician might be requested upon need. Initial therapy and clinical measurements: Following the screening examination, all subjects will receive a session of prophylaxis including instructions in proper oral hygiene measures. All clinical measurements at baseline and 6-months after surgery will be carried out by a calibrated examiner blinded to the provided treatment. Recession depth, and keratinized tissue height will be measured at the mid-buccal aspect of the treated tooth; probing depth, and clinical attachment level will be measured at the mesial, mid, and distal buccal/lingual aspect of the treated tooth; recession width will also be measured. Position of frenal attachment will be documented. All measurements will be performed by means of a PCP-15 manual periodontal probe and will be rounded up to the nearest millimeter. Recession depth will be measured as the distance between the cemento-enamel junction and gingival margin. Keratinized tissue height will be measured as the distance between the gingival margin and mucogingival junction. Intra-oral scanners will be used to capture scans at baseline and 6-months post-surgery. Randomization: Subjects will be assigned to one of the two treatment groups by blinded allocation. Randomization will be obtained with the use of computer-generated block randomization. The sealed envelope with treatment allocation will be assigned by the participant research number and opened at time of the surgery immediately before the treatment of the root surface. Surgical therapy: Under local anesthesia, a bilaminar (CAF+CTG) technique will be performed in the control group and a bilaminar (GPST+CTG) will be performed in the test group to accomplish root coverage. For CAF+CTG, in brief, exposed root surfaces will be mechanically treated with the use of curettes, a trapezoidal flap will be raised split/full thickness and a CTG will be sutured at the level of the cemento-enamel junction (CEJ). The flap will be coronally advanced and sutured with sling sutures anchored around the palatal cingulum of tooth with gingival recessions. For GPST+CTG, in brief, exposed root surfaces will be mechanically treated with the use of curettes. Starting from the line angle of the CEJ, a horizontal incision, whose length similar to the recession width, will be made distally or mesially. The distal point of the horizontal incision will be connected to a vertical incision which will be extended beyond the mucogingival junction (MGJ) and a split-thickness pedicle will be elevated. On the opposite side to the recession, a split-thickness tunnel will be prepared. CTG will be sutured at the level of CEJ with 1/3 of the length inserted into the prepared tunnel and the rest adapted to the recipient site. Finally, the pedicle will be rotated mesially to passively cover the middle portion of the graft and secured without tension. The CTG will be harvested from the palate using the single incision technique (Hurzeler and Weng 1999) or deepithelialized free gingival graft technique (Zucchelli et al 2010). The minimum thickness of CTG will be kept at 1.5 mm. Post-operative pain and edema will be controlled with ibuprofen 400 mg every 6-8 hours as needed. Patients will be instructed not to brush their teeth in the treated area but to rinse with chlorhexidine solution (0.12%) two times a day for 30 sec. for 6-weeks. Fourteen days after the surgical treatment, the sutures will be removed. Procedures done to ensure safety and minimize risks: The research team assembled have sufficient expertise and experience to conduct the research and will ensure that the projected sample size is sufficient to yield useful results. The surgical techniques being tested in this study are predictable procedures performed according to the current standards of care. The surgeries will be done by the residents of the Periodontics Department at CWRU, under strict supervision of a board-certified periodontist. Consequently, the delivery of standardized treatment of high quality will be ensured. In addition, the procedures will be performed conservatively with the aid of magnification and illumination to minimize the incidence of complications. The research team will meet regularly to evaluate the progress of the study, including periodic assessments of data quality and timelines, participant recruitment, accrual, and retention, and to ensure data integrity and confidentiality as well as adherence to the protocol

For subjects who learn about the study through advertisements or social media that express their interest in participation, pre-screening will be done through phone questionnaires prior to the actual informed consent/screening visit. Individuals who were deemed eligible in the pre-screening phase, as well as subjects recruited from the department of Periodontics at CWRU will be scheduled for an in-person visit. During this visit, they will be presented with the informed consent forms which will be thoroughly reviewed with each participant in an estimated time of one hour. Subjects who request a waiting period between being informed and consenting will be given a period of 48 hours. Upon consenting, screening will take place in the same visit. Screening will include gathering information such as demographics, medical history, clinical examination, and inclusion/exclusion criteria assessment. Prophylaxis will take place in the same visit and oral hygiene instructions will be reinforced. Recruitment will continue in the same manner and will be concluded upon completion of the sample size in an estimated period of 24 months. In the subsequent visit, surgeries will be performed according to the randomized allocation provided by the software. After 2 weeks, subjects will be asked to come for a 2-week follow-up for suture removal and outcome measurements. At 6 weeks and 6 months from the procedure, primary and secondary outcomes will be recorded again to enable comparing the changes from the baseline between the two surgical methods. The total timeline of the study is estimated to be around 36 months.

Sample size: The study is powered to detect a minimum clinically significant difference in root coverage of 1 mm using alpha = 0.05, a power = 80%, a hypothesized within-group sigma of 1 mm, obtained from previous studies. A total of 36 subjects will be recruited with an anticipated attrition of 20%. A minimum total of 30 subjects would be needed (15 test and 15 control) for an anticipated power of 84%. Proposed Analysis: The D'Agostino & Pearson normality test will be applied for each variable to test for normality. Descriptive statistics will be used for demographics while continuous variables will be tested for normal distribution using parametric tests such as paired T-test or two-group Analysis of Variance (ANOVA) with repeated measures, with follow-up Tukey's Honestly Significant Difference (HSD) tests as appropriate. Non-parametric data will be tested using Kruskal-Wallis or Mann Whitney U test.

ELIGIBILITY:
Inclusion Criteria:

* Males and females of > 18 years of age
* Single Cairo's RT1 (Recession Type 1) and RT2 ( Recession Type 2) recession defects (≥3 mm in depth) in mandibular anterior teeth (Incisors).
* Presence of identifiable cemento-enamel junction (CEJ)
* Presence of a step ≤1 mm at the CEJ level and/or the presence of a root abrasion, but with an identifiable CEJ, will be accepted
* Periodontally and systemically healthy patients
* No contraindications for periodontal surgery and not taking medications known to interfere with periodontal tissue health or healing; and no prior periodontal surgery on the involved sites

Exclusion Criteria:

* Vaping, chewing tobacco or smoking > 10 cigarettes per day
* Uncontrolled Diabetes Mellitus (HbA1c > 7)
* Pregnancy and Lactation
* Diseases affecting connective tissue metabolism
* Long-term steroid use
* Recession defects associated with caries
* Teeth associated with pulpal pathology

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-05-19 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of mean root coverage | 6 months
  The mean of the amount of root coverage will be calculated within and between test and control groups.

SECONDARY OUTCOMES:
Percentage of complete root coverage | 6 months
  The percentage of teeth that achieved complete root coverage will be compared between test and control.
Keratinized Tissue gain. | 6 months
  The changes in the amount of keratinized tissue from baseline to 6 months will calculated within and between study groups

CONTACTS AND LOCATIONS:
Overall Officials: Gian Pietro Schincaglia, DDS, PhD, Principal Investigator — Case Western Reserve University
Locations (1):
- Case Western Reserve University School of Dental Medicine, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No